CLINICAL TRIAL: NCT02999698
Title: A Comparative Retrospective Study Between Patients With Hidradenitis vs Patients With Psoriasis: Psychological Impact
Brief Title: Patients With Hidradenitis vs Patients With Psoriasis: Psychological Impact
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Universitat Autonoma de Barcelona (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-PSI-2016-71
Record Dates: First submitted 2016-12-19; First posted 2016-12-21 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Psoriasis; Hidradenitis
Keywords: Psoriasis; Hidradenitis; Psychological impact; Quality of life
MeSH Terms: conditions — Psoriasis; Hidradenitis | interventions — Watchful Waiting

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Psoriasis Group: Patients with psoriasis complete the questionnaires for psychological impact.
  Interventions: Other: Observational
- Hidradenitis Suppurativa Group: Patients with hidradenitis suppurativa complete the questionnaires for psychological impact.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Observational

SUMMARY:
The aim of this study is to evaluate the psychological impact of psoriasis or hidradenitis suppurativa on patients, in order to compare both pathologies.

ELIGIBILITY:
Inclusion Criteria:

* Men and women at least 18 years old at the time of selection.
* Subjects diagnosed with psoriasis or hidradenitis suppurativa
* Subjects who had completed the questionnaires for psychological impact.
* Patients should be able to understand and communicate with the investigator.

Exclusion Criteria:

* Subjects suffering from a serious concomitant illness.
* Subjects with a mental illness.
* Subjects who are performing psychiatric treatment.
* Patients who have alcohol dependence or drug abuse.
* Subjects that present legal incapacity or limited legal capacity.
* Subjects presenting illiteracy or language barriers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with hidradenitis suppurativa or psoriasis who have completed the questionnaires for psychological impact in the Hospital de la Santa Creu and Sant Pau, Barcelona.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-02; Primary Completion 2017-04 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Dermatology Quality of Life Index (DLQI) | 1 day
  The Dermatology Life Quality Index or DLQI, developed in 1994, was the first dermatology-specific Quality of Life instrument. It is a simple 10-question validated questionnaire that has been used in over 40 different skin conditions in over 80 countries and is available in over 90 languages. Its use has been described in over 1000 publications including many multinational studies. The DLQI is the most frequently used instrument in studies of randomised controlled trials in dermatology.
Hospital Anxiety and Depression Scale (HADS) | 1 day
  Hospital Anxiety and Depression Scale (HADS) was originally developed by Zigmond and Snaith (1983) and is commonly used by doctors to determine the levels of anxiety and depression that a patient is experiencing. The HADS is a fourteen item scale that generates ordinal data. Seven of the items relate to anxiety and seven relate to depression.
Perceived Stress Scale (PSS) | 1 day
  Perceived Stress Scale (PSS) was originally developed by Cohen (1983) and this scale is a self-report instrument that evaluates the level of stress perceived during the last month. The scale consists of 14 items with a response format of a five-point scale (0 = never, 1 = almost never, 2 = Every now and then, 3 = often, 4 = very often). The score obtained indicates that a higher score corresponds to a higher level of perceived stress.
The Holmes and Rahe stress scale | 1 day
  The Holmes and Rahe stress scale is a list of 43 stressful life events that can contribute to illness.

SECONDARY OUTCOMES:
Psoriasis Area Severity Index (PASI) | 1 day
  The Psoriasis Area Severity Index (PASI) is an index used to express the severity of psoriasis. It combines the severity (erythema, induration and desquamation) and percentage of affected area.
Static Physician's Global Assessment (sPGA) | 1 day
  The PGA is a 5 point ordinal rating ranging from "clear" to "very severe psoriasis".
Hurley's staging system | 1 day
  Hurley separated patients into three groups based largely on the presence and extent of cicatrization and sinuses. It has been used as a basis for clinical trials in the past and is a useful basis to approach therapy for patients. These three stages are based on Hurley's staging system, which is simple and relies on the subjective extent of the diseased tissue the patient has. Hurley's three stages of hidradenitis suppurativa.
Hidradenitis Suppurativa - Physician Global Assessment (HS-PGA) | 1 day
  The six-point Physician Global Assessment (PGA) ranges from clear to very severe. It is used in clinical trials to measure clinical improvement in inflammatory nodules, abscesses and draining fistulae

CONTACTS AND LOCATIONS:
Overall Officials: Esther Margarit de Miguel, Msc, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau; Antoni Font Guiteras, PhD, Study Director — Universitat Autonoma de Barcelona

IPD SHARING:
Plan to Share IPD: No